CLINICAL TRIAL: NCT02263144
Title: Resect and Discard Extension to Fuji Intelligent Color Enhancement (FICE) of Narrow Band Imaging International Colorectal Endoscopic (NicE) Classification
Brief Title: Resect and Discard Extension to FICE of NIcE Classification
Acronym: FICE;NICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Royal Alexandra Hospital (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Nuovo Regina Margherita Hospital (Other); University of Erlangen-Nürnberg Medical School (Other); University Hospital Regensburg (Other); Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Responsabile Progetto Ricerca Clinica, Istituto Clinico Humanitas
Other Study IDs: REDEFINE
Record Dates: First submitted 2014-09-25; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Hyperplastic Polyps; Adenomatous Polyps
MeSH Terms: conditions — Adenomatous Polyps

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — colonic polyps
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- histologically-verified <10mm polyps: histologically-verified <10mm polyps, analyzed by virtual chromo-endoscopy using FICE Fujifilm Technology
  Interventions: Procedure: virtual chromo-endoscopy using FICE Fujifilm Technology

INTERVENTIONS:
Procedure: virtual chromo-endoscopy using FICE Fujifilm Technology — For each polyps, any observer will use virtual chromo-endoscopy with FICE Fujifilm Technology

SUMMARY:
The purpose of this prospective, non-interventional study is to validate the Narrow Band Imaging International Colorectal Endoscopic (NICE) classification for differentiating subcentimetric hyperplastic and adenomatous polyps by using Fuji Intelligent Color Enhancement (FICE) technology with high-definition without optical magnification.

DETAILED DESCRIPTION:
1. In order to create a video-library of endoscopic cases, patients undergoing screening or diagnostic colonoscopy will be considered for inclusion. Patients with at least one histologically verified <10 mm polyp will be included. A short video-clip (around 15-20 seconds) of each polyp both at white-light and FICE-light will be recorded and stored in an anonymized database.
2. Once the video-library is completed, each of 7 experts will independently review all the cases. For each case, any observer will assess each of the three NICE criteria (colour/vascularization/surface), the degree of confidence (low/high), and classify the lesion as neoplastic or non-neoplastic. The primary outcomes are the accuracy of FICE technology with high-definition and without magnification, when adopting NICE classification, to differentiate between hyperplastic and adenomatous lesions, and the inter-observer agreement in such differentiation. Secondary end-points are to assess at multivariate measure the role of any individual criteria of NICE classification in the discrimination between the two histotypes, and possible adaptations of NICE classification in order to be applied with FICE.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is undergoing colonoscopy for screening, for surveillance in follow-up of previous polypectomy or for diagnostic work-up;
2. The patient is at satisfactory risk to undergo abdominal surgery;
3. The patient must understand and provide written consent for the procedure.

Exclusion Criteria:

1. Patients with inflammatory bowel disease;
2. Patients with a personal history of polyposis syndrome;
3. Patients with diverticulitis or toxic megacolon;
4. Patients with a history of radiation therapy to abdomen or pelvis.
5. Patients with a history of severe cardiovascular, pulmonary, liver or renal disease;
6. Personal history of coagulation disorders or use of anticoagulants
7. Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive adult patients who were referred for elective outpatient colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
accuracy of the NICE criteria using FICE technology for differentiating between the non-neoplastic and neoplastic histotypes in diagnoses with high-confidence on a video-library of 110 polyps reviewed by 7 experts. | up to 6 months
  7 experts will review videos from a video-library of subcentimetric polyps removed and histologically verified and will assess each of the three NICE criteria (colour/vascularization/surface), and classify the lesion as neoplastic or non-neoplastic with low or high confidence.
Inter-observer agreement among the 7 experts | up to 6 months
  The inter-observer agreement, among the 7 experts, on the final diagnosis (neoplastic or non-neoplastic) and on each individual NICE criterion for each polyp will be determined by using K statistics .

OTHER OUTCOMES:
Accuracy of additional criteria, such as the presence of mucus, to differentiate between sub-types of non-neoplastic lesions (i.e. serrated lesions) | up to 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (7):
- Dept of Gastroenterology and Endoscopy, University Hospital, Leuven, Belgium
- Dept of Gastroenterology, Edouard Herriot Hospital, Hospices Civils of Lyon, Lyon, France
- Germany (2):
  - Department of Medicine I, University of Erlangen-Nürnberg Medical School, Erlangen
  - Dept of Gastroenterology and interventional Endoscopy, Krankenhaus Barmherzige Brüder, Regensburg
- Italy (2):
  - Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano
  - Digestive Endoscopy Unit, Nuovo Regina Margherita Hospital, Rome
- Solent Centre for Digestive Diseases , Royal Alexandra Hospital, Portsmouth, United Kingdom

REFERENCES:
- [Background] Hewett DG, Kaltenbach T, Sano Y, Tanaka S, Saunders BP, Ponchon T, Soetikno R, Rex DK. Validation of a simple classification system for endoscopic diagnosis of small colorectal polyps using narrow-band imaging. Gastroenterology. 2012 Sep;143(3):599-607.e1. doi: 10.1053/j.gastro.2012.05.006. Epub 2012 May 15. PMID 22609383